CLINICAL TRIAL: NCT07034378
Title: Comparison of Extended Cryoballoon Ablation, Standard Cryoballoon Ablation, and Radiofrequency Catheter Ablation in Patients With Persistent Atrial Fibrillation: A Multicenter, Randomized Controlled Clinical Trial
Brief Title: Comparison Between Extended Cryoablation, Standard Cryoablation, and Radiofrequency Ablation
Acronym: EXCAPE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Gi-Byoung Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2020-1896
Record Dates: First submitted 2025-05-12; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Extended cryoballoon ablation (Experimental): The method of ablation, size of balloon, freezing time, and booster freezing will be decided by the participating center's policy or physician's discretion. Ablation strategies described above are highly recommended for all participants.
  Additional posterior wall isolation should be performed by single 120 to 180 second CB application delivered at each site. Maximal posterior wall debulking should be attempted, although complete isolation may not always be achievable, as we considered that a large scar created by the CB application would provide sufficient anti-arrhythmic effects in terms of suppressing AF. The number and duration of CB application should be recorded in the case report form. Successful posterior wall isolation should be determined by 3-dimensional electro-anatomical mapping or differential pacing. The method and achievement of posterior wall isolation should be recorded in the case report form.
  Interventions: Procedure: Extended cryoballoon ablation
- Standard cryoballoon ablation (Active Comparator): Application of TTI + 2 minutes or 180 seconds single-freezing is recommended when time-to-isolation (TTI) <60 seconds. Additional 120 seconds of booster-freezing after TTI + 2 or 180 seconds initial freezing is recommended when TTI value >60 seconds, or PV potentials were not discernable in the Achieve multipolar catheter. If temperatures below -40°C cannot be achieved due to improper occlusion or TTI > 90 seconds, freezing should be discontinued and reposition of balloon is recommended. Segmental ablation is allowed when the proper occlusion of PV by balloon cannot be achieved. Continuous phrenic capture should be monitored during the procedure in the right PVs to avoid phrenic nerve injury. Stop ablation immediately if phrenic nerve damage is suspected. No further ablation would be performed if the phrenic nerve damage is suspected. Touch-up ablation using irrigated radiofrequency ablation catheter would be permitted with conventional mapping method.
  Interventions: Procedure: Standard cryoballoon ablation
- Radiofrequency ablation (Active Comparator): CARTO system (Biosense-Webster, USA): Ablation index (AI) CLOSE protocol . Navistar Smart-touch surround-flow catheter; 25-40 watts of energy; 40 seconds time limit; 10-30 gram of contact force; 40 seconds time limit; targeting AI value of 550 in anterior wall and 400 in the posterior wall; interlesion distance ≤6mm; using automatic lesion annotation (Visitag™) - type 3 tagging, 3mm stability for 5 seconds, force >5g over 50% of time; target AI value could be reduced (450 in anterior wall and 350 in posterior wall) according to the participating center's policy.
  Ensite NavX system (Abbott, USA) :
  TactiCath™ Quartz ablation catheter; delivering 25-35 watts of energy; 40 seconds time limit; 10-30 gram of contact force; using automatic lesion annotation (Automark Module), target lesion index value of 5-5.5 in the posterior wall and 5.5-6 in the anterior wall.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation of pulmonary veins
  Arms: Radiofrequency ablation
Procedure: Extended cryoballoon ablation — Cryoablation of pulmonary veins + posterior wall isolation
  Arms: Extended cryoballoon ablation
Procedure: Standard cryoballoon ablation — Standard cryoablation of pulmonary veins
  Arms: Standard cryoballoon ablation

SUMMARY:
The objective of this study is to test the efficacy hypothesis that extended cryoballoon ablation is superior to either standard cryoballoon ablation or radiofrequency ablation

DETAILED DESCRIPTION:
The posterior wall of the left atrium is known to contribute to arrhythmogenicity and has been associated with higher rates of atrial fibrillation (AF) recurrence. In this trial, we aim to evaluate whether extended cryoballoon ablation-comprising pulmonary vein isolation (PVI) plus posterior wall isolation-results in superior rhythm outcomes compared to standard cryoballoon ablation (PVI only) or radiofrequency ablation (PVI only). Patients will be randomly assigned to one of three treatment arms: extended cryoballoon ablation, standard cryoballoon ablation, or radiofrequency ablation. Each patient will receive the assigned treatment accordingly. The primary outcome is the incidence of atrial tachyarrhythmias-including atrial fibrillation, atrial flutter, and atrial tachycardia-lasting more than 30 seconds, occurring after discontinuation of antiarrhythmic drugs and following a 3-month post-procedure blanking period. Outcomes will be compared at 1 year after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-80 years
* Patients with persistent (≥7 days) AF documented on 12-lead ECG or Holter monitoring.
* AF refractory/intolerant to class I or III antiarrhythmic drugs
* Able and willing to provide written informed consent to CB or RF ablation and participation in this investigation

Exclusion Criteria:

* Age <18 years old or >80 years old
* Paroxysmal AF lasting <7 days
* Mitral stenosis or mechanical prosthetic valve
* Patients with left atrial size ≥ 50 mm (2D echocardiography, Anterior-posterior diameter in parasternal long axis view)
* Anatomy of pulmonary vein not suitable for standard CB or extended CB, including common ostium or ostium size > 26mm
* Pregnant woman of childbearing age with a positive pregnancy test before treatment
* Presence of atrial septal defect or patent foramen ovale closure device
* Presence of intracardiac thrombus
* Contraindications to the systemic anticoagulation
* NYHA functional class IV heart failure
* Prior catheter or surgical ablation of AF
* Acute coronary syndrome within 3 months
* Planned open heart surgery within 3 months
* Prior open-heart surgery within 3 months
* End stage renal disease or chronic kidney disease (estimated glomerular filtration rate [MDRD method] < 30mL/min/1.73m²)
* Life expectancy less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
the incidence rates of atrial tachyarrhythmias | 3-month blanking period post-procedure
  Incidence of atrial tachyarrhythmias (including atrial fibrillation, flutter, or tachycardia) lasting >30 seconds after discontinuation of antiarrhythmic therapy, assessed following a 3-month blanking period

SECONDARY OUTCOMES:
Atrial arrhythmia recurrence during blanking period | during blanking period (3 months)
  Atrial arrhythmia recurrence during blanking period (3 months) after one or two procedures with/without antiarrhythmic medications
Atrial tachycardia or flutter recurrence | 1 year
  Atrial tachycardia or flutter recurrence during long-term follow-up after one or two procedures with/without antiarrhythmic medications
Atrial fibrillation recurrence | 1 year
  Atrial fibrillation recurrence during long-term follow-up after one or two procedures with/without antiarrhythmic medications
Incidence of peri-procedural complications | Periprocedural
  including stroke, cardiac tamponade, esophageal injury, phrenic nerve damage, and death
Rate of first-pass isolation or first-freeze isolation | during procedure
Procedure duration (minutes) | during procedure
Ablation time (minutes) | during procedure
Fluoroscopy time (minutes) | during procedure
LA dwelling time | during procedure
Ablation time (seconds) | during procedure
Quality of life changes at 12 months compared to baseline | 1 year
  Scores from the SF-36 questionnaire will be compared between baseline and the 1-year follow-up period. Scores will be scaled from 0 to 100, with higher values indicating better quality of life
Number of repeat procedures | 1 year
AF burden by 2-week patch monitoring | 1 year
  AF burden assessed at 12 months after ablation
LA pressure, mmHg (max/min/mean) | during procedure

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No